CLINICAL TRIAL: NCT00708994
Title: Cannabinoids, Psychosis, Neural Synchrony, and Information Processing
Brief Title: Cannabinoids, Neural Synchrony, and Information Processing
Acronym: THC-Gamma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Associate Professor, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0803003638; 5R21DA020750-02 (NIH)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Cannabis; Psychotic Disorders
MeSH Terms: conditions — Marijuana Abuse; Psychotic Disorders | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- THC (Active Comparator): * Very low dose (0.0015 mg/kg = 0.21 mg in a 70kg individual) THC, dissolved in alcohol. Administered intravenously over 10 minutes.
  * Low dose (0.015 mg/kg = 1.05 mg in a 70kg individual) THC, dissolved in alcohol. This dose is roughly equivalent to smoking approximately 1/4th of a marijuana cigarette, or "joint". Administered intravenously over 10 minutes.
  * Medium dose (0.03 mg/kg = 2.1 mg in a 70 kg individual) THC, dissolved in alcohol. This dose is roughly equivalent to smoking approximately 1/2 of a marijuana cigarette, or "joint". Administered intravenously over 10 minutes.
  Interventions: Drug: THC
- Placebo (Placebo Comparator): • Control: small amount of alcohol intravenous (quarter teaspoon), with no THC over 10 minutes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THC — * Very low dose (0.0015 mg/kg = 0.21 mg in a 70kg individual) THC, dissolved in alcohol. Administered intravenously over 10 minutes.
  * Low dose (0.015 mg/kg = 1.05 mg in a 70kg individual) THC, dissolved in alcohol. This dose is roughly equivalent to smoking approximately 1/4th of a marijuana cigarette, or "joint". Administered intravenously over 10 minutes.
  * Medium dose (0.03 mg/kg = 2.1 mg in a 70 kg individual) THC, dissolved in alcohol. This dose is roughly equivalent to smoking approximately 1/2 of a marijuana cigarette, or "joint". Administered intravenously over 10 minutes.
  Arms: THC
Drug: Placebo — • Control: small amount of alcohol intravenous (quarter teaspoon), with no THC over 10 minutes
  Arms: Placebo

SUMMARY:
The study examines the effects of delta-9-tetrahydrocannabinol (Δ9-THC), the principal active ingredient of cannabis, on neural synchrony. Neural synchrony is studied using electroencephalography (EEG).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and 55 years (extremes included) on the day of the first dosing.
* Exposed to cannabis at least once.

Exclusion Criteria:

1. Cannabis naïve
2. Positive pregnancy screen during screening
3. Hearing deficits

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2008-02-25 (Actual); Primary Completion 2012-12-03 (Actual); Study Completion 2012-12-03 (Actual)

PRIMARY OUTCOMES:
EEG | +30
Clinician Administered Dissociative Symptoms Scale, Positive and Negative Symptom Scale, Visual Analog Scale | Baseline, +10, +80

CONTACTS AND LOCATIONS:
Overall Officials: Deepak D'Souza, MD, Principal Investigator — Yale University Medical School
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Ranganathan M, Radhakrishnan R, Addy PH, Schnakenberg-Martin AM, Williams AH, Carbuto M, Elander J, Pittman B, Andrew Sewell R, Skosnik PD, D'Souza DC. Tetrahydrocannabinol (THC) impairs encoding but not retrieval of verbal information. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Oct 3;79(Pt B):176-183. doi: 10.1016/j.pnpbp.2017.06.019. Epub 2017 Jun 20. PMID 28642081